CLINICAL TRIAL: NCT05902234
Title: Emotional Bodymaps in Pediatric Pain Patients and Their Parents.
Acronym: PedPainEmot
Status: Recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Reetta Sipilä, PhD, Helsinki University Central Hospital
Other Study IDs: HUS/1301/2023
Record Dates: First submitted 2023-05-23; First posted 2023-06-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric pain patients and their parents: patients and their parents
  Interventions: Behavioral: interdiciplinary treatment

INTERVENTIONS:
Behavioral: interdiciplinary treatment — Normal interdiciplinary treatment path

SUMMARY:
The aims of this study are to find out how pain may alter the experience of emotions in the body in pediatric pain patients and how how their parent feel the emotions in their bodies. We are also interested how this possible effect is mediated by the duration and location of pain, mood changes or with the experience of bullying.

ELIGIBILITY:
Inclusion Criteria:

* fluency in finnish language

Exclusion Criteria:

* none

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pediatric pain clinic patients and their parents
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
emotional bodymaps | 10months
  sensations of emotion in ones body

SECONDARY OUTCOMES:
pain PROMIS | 10 months
  pain interference and intensity
psychological flexibility | 10 months
  measure of psychological flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Reetta M Sipilä, PhD, Principal Investigator — HUS, HY
Locations (1):
- New Childrens Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided